CLINICAL TRIAL: NCT03543865
Title: Southwest Hub for American Indian Youth Suicide Prevention Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB00008138-2; 5U19MH113136-02 (NIH); NCT03132766 (obsolete NCT alias)
Record Dates: First submitted 2018-04-13; First posted 2018-06-01 (Actual); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Suicide; Surveillance; Mental Health; Substance Use; Depressive Symptoms
Keywords: American Indian; Resilience; Native American
MeSH Terms: conditions — Suicide; Psychological Well-Being; Substance-Related Disorders; Depression | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- New Hope (NH) (Experimental): The investigators will employ a SMART design to evaluate the effectiveness of New Hope (NH), Elders' Resilience intervention (ER), Case Management (CM) and the combination of these approaches on reducing suicidal thoughts and promoting resilience among AI youth ages 10-29 who are confirmed by surveillance case managers to have recently experienced suicide ideation, attempt or a binge substance use and ideation.
  Youth who assent will complete the baseline (CM visit 1 and will be referred to mental health care). During the same visit, youth will be randomized 1:1 to either New Hope (NH) plus Case Management (CM), or CM alone, using a blocked randomized design, stratifying participants by age and event type.
  Interventions: Behavioral: New Hope (NH); Other: Case Management (CM)
- Elders' Resiliency (ER) (Experimental): The investigators will employ a SMART design to evaluate the effectiveness of New Hope (NH), Elders' Resilience intervention (ER), Case Management (CM) and the combination of these approaches on reducing suicidal thoughts and promoting resilience among AI youth ages 10-29 who are confirmed by surveillance case managers to have recently experienced suicide ideation, attempt or a binge substance use and ideation.
  All youth will complete another study assessment after 30 days. The 30-day time frame will allow ample time to complete the NH intervention with participants and assess any changes in youth's mental health status for all study arms. Following another 30-day period, all participants will be re-assessed and re-randomized, using the same blocking and 1:1 ratio to either the Elders' Resilience (ER) intervention plus CM, or CM alone. To track long term outcomes, all youth will complete a final assessment 3 month later (6 months post-enrollment).
  Interventions: Behavioral: Elders Resilience (ER); Other: Case Management (CM)
- Control Condition (Other): The control condition will only receive Case Management (CM) (n=76).
  The investigators will employ a SMART design to evaluate the effectiveness of New Hope (NH), Elders' Resilience intervention (ER), Case Management (CM) and the combination of these approaches on reducing suicidal thoughts and promoting resilience among AI youth ages 10-29 who are confirmed by surveillance case managers to have recently experienced suicide ideation, attempt or a binge substance use and ideation. Youth who assent will complete the baseline (CM visit 1 and will be referred to mental health care). During the same visit, youth will be randomized 1:1 to either New Hope (NH) plus Case Management (CM), or CM alone, using a blocked randomized design, stratifying participants by age and event type.
  Interventions: Other: Case Management (CM)
- New Hope (NH), Elders' Resiliency (ER), Case Management (CM) (Experimental): The investigators will employ a SMART design to evaluate the effectiveness of New Hope (NH), Elders' Resilience intervention (ER), Case Management (CM) and the combination of these approaches on reducing suicidal thoughts and promoting resilience among AI youth ages 10-29 who are confirmed by surveillance case managers to have recently experienced suicide ideation, attempt or a binge substance use and ideation. Youth who assent will complete the baseline (CM visit 1 and will be referred to mental health care). During the same visit, youth will be randomized 1:1 to either New Hope (NH) plus Case Management (CM), or CM alone, using a blocked randomized design, stratifying participants by age and event type. All youth will complete another study assessment after 30 days.After another 30-days, all participants will be re-assessed/re-randomized, using the same blocking and 1:1 ratio to either the ER intervention plus CM, or CM alone.
  Interventions: Behavioral: New Hope (NH); Behavioral: Elders Resilience (ER); Other: Case Management (CM)

INTERVENTIONS:
Behavioral: New Hope (NH) — New Hope will be implemented over 1 visit (2-4 hours) in a youth-preferred setting after Emergency Department (ED) discharge for a suicide attempt, and in the past few years has been updated to also target suicide ideation and binge behavior. NH emphasizes the seriousness of a suicide attempt; teaches coping skills to reduce risk, including emotion regulation, cognitive restructuring, social support, and safety planning; and helps participants overcome barriers to treatment motivation, initiation, and adherence. A center-piece of the intervention is a 20-minute video produced by with Native actors, vignettes specific to this community, and Elders speaking in Apache (with sub-titles) about the seriousness of suicide, its impact on the community, their concern for the adolescent, and beliefs about the communal importance of each individual's life.Youth will be encouraged to choose a support person from his/her family to take part in the intervention.
  Arms: New Hope (NH); New Hope (NH), Elders' Resiliency (ER), Case Management (CM)
Behavioral: Elders Resilience (ER) — Elders' Resiliency is a monthly manualized curriculum taught by Elders in the community intended to bolster Apache youths' resilience to suicide ideation, attempts and substance abuse by promoting Apache cultural identity and values, youth's self-worth and role in the community, and fostering connectedness to society and community, with an emphasis on extended family as a nexus of strength. Each lesson introduces youth to cultural knowledge, stories, and songs with an emphasis on respect and the sacredness of each life. Our community-based Apache staff will select Elders who both express an interest in the current project and have demonstrated affinity and skill for teaching the current curriculum in the schools. After this group of Elders is recruited and agree to participate, they will be paired with our paraprofessional Apache study staff.
  Arms: Elders' Resiliency (ER); New Hope (NH), Elders' Resiliency (ER), Case Management (CM)
Other: Case Management (CM) — Research Program Assistants, who are trained Surveillance System Staff, will conduct the monitoring and case management visits in participants' homes or other private settings at baseline, 1, 2, 3 and 6 months post-enrollment. The CM visit includes rapport-building, use of the Suicide Ideation Questionnaire (SIQ) to assess imminent risk, and if youth report not yet having connected to services, referral to Apache Behavioral Health Services (ABHS), the local community mental health center. At CM visits, the Research Program Assistants will also monitor participants' completion of the study battery, which will be self-administered using tablets. In addition, Research Program Assistants will score the SIQ before leaving the youth. If the SIQ reveals the participant is at imminent risk, Research Program Assistants will employ a protocol for rescue services, which involves triaging youth immediately to the ED for further assessment and care.

SUMMARY:
1. To use a SMART design to evaluate which of four sequences of New Hope (NH), Elders Resilience (ER) and Case Management (CM) have the greater effects on immediate and longer-term suicidal ideation (primary outcome) and resilience (secondary outcome) among American Indian (AI) adolescents ages 10-29 identified at risk for suicide.

   Hypotheses:

   i. New Hope vs. CM alone will significantly reduce participant suicidal ideation.

   ii. Elders Resilience vs. CM alone will significantly improve participant resilience.

   iii. New Hope followed by Elders Resilience will have the strongest effects on suicidal ideation and resilience.

   iv. CM alone will have the weakest effects of all combinations.

   Secondary Aims:
2. To examine mediators and moderators of treatment effectiveness and sequencing in order to determine which types and sequence of interventions is best suited for which youth.
3. To assess the acceptability, feasibility and capacity for sustainability of the Hub's key intervention components (Surveillance/Case Management, New Hope and Elders' Resilience) from the perspective of multiple stakeholders as they are implemented across different tribes.

DETAILED DESCRIPTION:
The overall goal of the research component of the National Institute of Mental Health funded Southwest Hub for American Indian Youth Suicide Prevention Research is to identify effective, feasible and sustainable interventions to prevent suicide and promote resilience among American Indian (AI) youth. The proposed study will build on 20+ years of behavioral and mental health research and partnerships undertaken by the Center for American Indian Health (CAIH) at Johns Hopkins with the White Mountain Apache Tribe (WMAT).

The investigators primary research aim, to be undertaken with the White Mountain Apache, includes: 1) identification and voluntary enrollment of youth 10-29 years old using the WMAT established surveillance and case-management (CM) system who recently had a validated suicide attempt, ideation, or binge substance use episode with recent suicidal ideation; and 2) implementation of a Sequential Multiple Assignment Randomized Trial (SMART) to inform how to combine and tailor two brief interventions delivered by paraprofessional community mental health workers (CMHWs), with promising pilot data, to prevent further suicidal thoughts and behavior and promote resilience; and 3) evaluate what are the cost savings per study participant with the implementation of the Southwest Hub interventions: NH, ER, NH and ER. A secondary aim will be to evaluate the acceptability, feasibility and sustainability of the two brief interventions with other Southwest Hub partners, including the Navajo, San Carlos Apache, Hualapai, and Cherokee nations, who will have support from the Administrative Core of the Southwest Hub to implement their own local tribal suicide surveillance systems for community-based identification of at-risk youth.

The investigators will employ a SMART design to evaluate the effectiveness of New Hope (NH), Elders' Resilience intervention (ER), Case Management (CM) and the combination of these approaches on reducing suicidal thoughts and promoting resilience among AI youth ages 10-29 who are confirmed by surveillance case managers to have recently experienced suicide ideation, attempt or a binge substance use and ideation. Youth who assent will complete the baseline (case management visit 1 and will be referred to mental health care-the standard protocol for the Apache system). During the same visit, youth will be randomized 1:1 to either New Hope (NH) plus Case Management (CM), or CM alone, using a blocked randomized design, stratifying participants by age and event type. All youth will complete another study assessment after 30 days. The 30-day time frame will allow ample time to complete the NH intervention with participants and assess any changes in youth's mental health status for all study arms. Following another 30-day period, all participants will be re-assessed and re-randomized, using the same blocking and 1:1 ratio to either the Elders' Resilience (ER) intervention plus CM, or CM alone. To track long term outcomes, all youth will complete a final assessment 3 month later (6 months post-enrollment). This study will occur on the White Mountain Apache Tribe's Fort Apache reservation.

ELIGIBILITY:
Aim 1

Inclusion Criteria:

* Native American youth ages 10 to 29 years old.
* Reside on or near the Fort Apache Indian Reservation.
* Parent/guardian consent for youth under 18 years old.
* Suicide ideation, binge substance use with recent (i.e. within the last 3 months) suicide ideation, or suicide attempt in the past 30 days as identified and verified by the surveillance system or release from inpatient care related to suicide ideation or attempt within past 30 days.

Terms and Definitions: Definitions for reportable behaviors are modeled on the Columbia Classification Algorithm for Suicide Assessment (C- CASA).[11] Suicide attempt: intentional self-injury with intent to die. (Aborted and interrupted suicide attempts are included as part of this category). Suicidal ideation: thoughts to take one's own life with or without preparatory action. Binge substance use with recent ideation, defined by Apache stakeholders, as consuming substances with the intention of modifying consciousness and resulting in being found unresponsive or requiring ED treatment and answering positively to a 1-item screening question on the assessment indicating suicide ideation within the past three months.

Exclusion Criteria:

• Factors identified at baseline that preclude full participation, including: unstable and severe medical, psychiatric or drug use problem that necessitates inpatient treatment; acute suicidal or homicidal ideation requiring immediate intervention; recent, severe stressful life events such as physical or sexual abuse, or violent crime victimization that requires specific and high intensity interventions or out of home placement. Participants must speak English and not be severely visually impaired. Foster children will not be included. Ambiguous cases will be reviewed by one of the co-PIs before being deemed eligible for recruitment.

Aim 3

Inclusion Criteria:

* Youth over the age of 16 or adults over the age of 18.
* A person with an interest or concern related to youth suicide among AI populations.

Exclusion Criteria:

• Factors identified at baseline that preclude full participation including: being under the influence of a substance; active psychosis or mania; any other condition that makes an individual lack capacity to give consent. Foster children will not be included. Participants must speak English and not be severely visually impaired. Ambiguous cases will be reviewed by one of the co-PIs before being deemed eligible for recruitment.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 304 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Cwik, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for American Indian Health, Whiteriver, Arizona, United States

REFERENCES:
- [Derived] O'Keefe VM, Haroz EE, Goklish N, Ivanich J; Celebrating Life Team; Cwik MF, Barlow A. Employing a sequential multiple assignment randomized trial (SMART) to evaluate the impact of brief risk and protective factor prevention interventions for American Indian Youth Suicide. BMC Public Health. 2019 Dec 12;19(1):1675. doi: 10.1186/s12889-019-7996-2. PMID 31830933

RESULTS

PARTICIPANT FLOW:
Recruitment Details: N=304 participants were consented, N=284 completed baseline
Pre-assignment Details: N=284 participants completed baseline data and were randomized to the study arms. The participants who were not randomized were marked lost to follow-up if staff could not contact them further, or withdrawn if they requested to withdraw from the study.
Groups:
- New Hope (NH): Participants Receive New Hope and Case Management
- Elders' Resilience (ER): Participants Receive Elders' Resilience Curriculum and Case Management
- New Hope (NH) + Elders' Resilience (ER) + Case Management: Participants Receive New Hope, Elders' Resilience Curriculum and Case Management
- Case Management (CM): Case Management alone
Period: Overall Study
Arm/Group | New Hope (NH) | Elders' Resilience (ER) | New Hope (NH) + Elders' Resilience (ER) + Case Management | Case Management (CM)
Started | 71 | 68 | 65 | 80
Completed | 71 | 68 | 65 | 80
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- New Hope (NH): The investigators will employ a SMART design to evaluate the effectiveness of New Hope (NH), Elders' Resilience intervention (ER), Case Management (CM) and the combination of these approaches on reducing suicidal thoughts and promoting resilience among AI youth ages 10-24 who are confirmed by surveillance case managers to have recently experienced suicide ideation, attempt or a binge substance use and ideation.
  Youth who assent will complete the baseline (CM visit 1 and will be referred to mental health care). During the same visit, youth will be randomized 1:1 to either New Hope (NH) plus Case Management (CM), or CM alone, using a blocked randomized design, stratifying participants by age and event type.
- Elders' Resiliency (ER): The investigators will employ a SMART design to evaluate the effectiveness of New Hope (NH), Elders' Resilience intervention (ER), Case Management (CM) and the combination of these approaches on reducing suicidal thoughts and promoting resilience among AI youth ages 10-24 who are confirmed by surveillance case managers to have recently experienced suicide ideation, attempt or a binge substance use and ideation.
  All youth will complete another study assessment after 30 days. The 30-day time frame will allow ample time to complete the NH intervention with participants and assess any changes in youth's mental health status for all study arms. Following another 30-day period, all participants will be re-assessed and re-randomized, using the same blocking and 1:1 ratio to either the Elders' Resilience (ER) intervention plus CM, or CM alone. To track long term outcomes, all youth will complete a final assessment 3 month later (6 months post-enrollment).
- New Hope (NH), Elders' Resiliency (ER), Case Management (CM): The investigators will employ a SMART design to evaluate the effectiveness of New Hope (NH), Elders' Resilience intervention (ER), Case Management (CM) and the combination of these approaches on reducing suicidal thoughts and promoting resilience among AI youth ages 10-24 who are confirmed by surveillance case managers to have recently experienced suicide ideation, attempt or a binge substance use and ideation. Youth who assent will complete the baseline (CM visit 1 and will be referred to mental health care). During the same visit, youth will be randomized 1:1 to either New Hope (NH) plus Case Management (CM), or CM alone, using a blocked randomized design, stratifying participants by age and event type. All youth will complete another study assessment after 30 days.After another 30-days, all participants will be re-assessed/re-randomized, using the same blocking and 1:1 ratio to either the ER intervention plus CM, or CM alone.
- Control Condition: The control condition will only receive Case Management (CM) (n=76).
  The investigators will employ a SMART design to evaluate the effectiveness of New Hope (NH), Elders' Resilience intervention (ER), Case Management (CM) and the combination of these approaches on reducing suicidal thoughts and promoting resilience among AI youth ages 10-24 who are confirmed by surveillance case managers to have recently experienced suicide ideation, attempt or a binge substance use and ideation. Youth who assent will complete the baseline (CM visit 1 and will be referred to mental health care). During the same visit, youth will be randomized 1:1 to either New Hope (NH) plus Case Management (CM), or CM alone, using a blocked randomized design, stratifying participants by age and event type.
- Total: Total of all reporting groups
Arm/Group | New Hope (NH) | Elders' Resiliency (ER) | New Hope (NH), Elders' Resiliency (ER), Case Management (CM) | Control Condition | Total
Number analyzed (Participants) | 71 | 68 | 65 | 80 | 284
Age, Customized [Count of Participants; unit: Participants]
  Age: 14 and younger | 33 | 30 | 33 | 36 | 132
  Age: 15-19 | 19 | 17 | 20 | 28 | 84
  Age: 20-24 | 12 | 18 | 10 | 12 | 52
  Age: 25-29 | 7 | 3 | 2 | 4 | 16
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 19 | 20 | 12 | 21 | 72
  Sex: Female | 51 | 48 | 51 | 59 | 209
  Sex: Do not wish to disclose | 0 | 0 | 1 | 0 | 1
  Sex: Missing | 1 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 71 | 68 | 65 | 80 | 284
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Centers for Epidemiologic Studies of Depression (CESDR-10)
Description: The Centers for Epidemiologic Studies of Depression (CESDR-10) is a self-report scale used to measure depressive symptoms (Cronbach's alpha ranged from 0.90 to 0.91 in a validation study). Scores on the CESDR-10 range from 0 (minimum) to 40 (maximum) with higher scores representing higher frequency of experiencing depression symptoms. CESDR-10 score is summed to provide an overall total for each participant. The full version has been widely used among adolescent and AI populations, including Apache youth.
Time Frame: Baseline, 30 days, 60 days, 90 days, 180 days
Population: Participants with data collected
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | New Hope (NH) | Elders' Resiliency (ER) | Control Condition | New Hope (NH), Elders' Resiliency (ER), Case Management (CM)
Number analyzed (Participants) | 71 | 68 | 80 | 65
score on a scale
  Baseline | 15 [7 to 23] | 15 [5.5 to 21] | 14.5 [8 to 20] | 11 [5 to 24]
  30 Days: number analyzed (Participants) | 30 | 55 | 63 | 44
  30 Days | 8 [0 to 18] | 12 [4 to 18] | 13 [6 to 20] | 8 [2 to 19]
  60 Days: number analyzed (Participants) | 43 | 57 | 57 | 49
  60 Days | 7 [0 to 19] | 11 [3 to 18] | 9 [4 to 16] | 6 [1 to 17.5]
  90 Days: number analyzed (Participants) | 39 | 37 | 63 | 42
  90 Days | 9.5 [1 to 19] | 11.5 [5.5 to 17] | 8 [3 to 18] | 5.5 [2 to 17]
  180 Days: number analyzed (Participants) | 52 | 52 | 70 | 57
  180 Days | 4 [2 to 14] | 8.5 [2.5 to 15.5] | 6 [0 to 13] | 5.5 [1 to 13.5]

2. Secondary Outcome: The Children's Hope Scale (CHS)
Description: Children's Hope Scale, a 6-item measure assessing goal-directed thinking and pathways to achieve goals. Items are rated on a 6-point Likert scale (0=None of the time to 5=All of the time).
  Scoring Method: The total Hope Score is calculated by summing all 6 items. Score Range: 0 to 30
  Interpretation:
  * Higher scores indicate greater hope (better outcome)
  * Lower scores indicate lower hope (worse outcome)
Time Frame: Baseline, 30 days, 60 days, 90 days, 180 days
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Hope (NH) | Elders' Resiliency (ER) | Control Condition | New Hope (NH), Elders' Resiliency (ER), Case Management (CM)
Number analyzed (Participants) | 71 | 68 | 80 | 65
units on a scale
  Baseline | 14.4 (7.9) | 14.2 (7) | 15.2 (7.7) | 14.6 (7.5)
  30 Days: number analyzed (Participants) | 30 | 55 | 63 | 44
  30 Days | 17.6 (8.8) | 13.5 (7.3) | 15.2 (8.4) | 16.8 (8.2)
  60 Days: number analyzed (Participants) | 43 | 57 | 57 | 49
  60 Days | 16.4 (8.9) | 15.2 (8.2) | 17.6 (7.3) | 15.8 (8.5)
  90 Days: number analyzed (Participants) | 39 | 37 | 63 | 42
  90 Days | 17 (8.4) | 15.8 (8.2) | 18.7 (7.9) | 17.2 (8.7)
  180 Days: number analyzed (Participants) | 52 | 52 | 70 | 57
  180 Days | 18.2 (8) | 18.4 (7.2) | 18.4 (8.3) | 18.7 (8.1)

3. Secondary Outcome: Multicultural Mastery Scale
Description: Multicultural Mastery Scale, an adapted version measuring problem-solving through social networks across three domains: Mastery-Friends (4 items), Mastery-Family (4 items), and Mastery-Self (5 items), totaling 13 items.
  Items were assessed using either a slider scale (0-100) recoded to a 5-point scale, or a 3-point scale (0=Not at all, 1=Somewhat, 2=A lot) rescaled to a 5-point format. The final scoring uses a 5-point scale where each item ranges from 0 to 4.
  Scoring Method: The total Communal Mastery Score is calculated by summing all 13 items.
  Score Range: 0 to 52
  Interpretation:
  * Higher scores indicate a stronger sense of mastery and control (better outcome)
  * Lower scores indicate lower mastery (worse outcome)
Time Frame: Baseline, 30 days, 60 days, 90 days, 180 days
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Hope (NH) | Elders' Resiliency (ER) | Control Condition | New Hope (NH), Elders' Resiliency (ER), Case Management (CM)
Number analyzed (Participants) | 71 | 68 | 80 | 65
units on a scale
  Baseline | 30.7 (11.5) | 29.9 (10) | 30.7 (11.8) | 30.9 (10.0)
  30 Days: number analyzed (Participants) | 30 | 55 | 63 | 44
  30 Days | 34.2 (11.2) | 29 (9.9) | 29 (13.2) | 33 (10.5)
  60 Days: number analyzed (Participants) | 43 | 57 | 57 | 49
  60 Days | 32.2 (13.1) | 30.6 (11.7) | 35.2 (9.2) | 29.8 (11)
  90 Days: number analyzed (Participants) | 39 | 37 | 63 | 42
  90 Days | 32.7 (11.4) | 31 (8.4) | 33.9 (10.6) | 30.3 (13.4)
  180 Days: number analyzed (Participants) | 52 | 52 | 70 | 57
  180 Days | 31.7 (9.6) | 32.7 (11.1) | 33.4 (11.2) | 35.8 (11.5)

4. Secondary Outcome: Rosenberg Self Esteem Scale
Description: The scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.
Time Frame: Baseline, 30 days, 60 days, 90 days, 180 days
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | New Hope (NH) | Elders' Resiliency (ER) | Control Condition | New Hope (NH), Elders' Resiliency (ER), Case Management (CM)
Number analyzed (Participants) | 71 | 68 | 80 | 65
score on a scale
  Baseline | 17.5 (3.7) | 17.7 (3.9) | 17.5 (3.5) | 16.5 (4.9)
  30 Days: number analyzed (Participants) | 30 | 55 | 63 | 44
  30 Days | 15.8 (4.1) | 16.5 (4.2) | 16.5 (5.3) | 17.2 (3.1)
  60 Days: number analyzed (Participants) | 43 | 57 | 57 | 49
  60 Days | 15.9 (5.6) | 17.3 (3.4) | 18.1 (4.7) | 17.5 (4.8)
  90 Days: number analyzed (Participants) | 39 | 37 | 63 | 42
  90 Days | 16.6 (3.8) | 16.5 (5.8) | 17.8 (4.5) | 16.5 (5.8)
  180 Days: number analyzed (Participants) | 52 | 52 | 70 | 57
  180 Days | 16.8 (3.6) | 17.4 (4.2) | 16.8 (5.4) | 16.1 (4.9)

5. Secondary Outcome: Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) Risk Score
Description: The World Health Organization (WHO) Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) is a questionnaire that screens for all levels of problem or risky substance use in adults. A risk score can be provided for each substance, and scores are grouped into low risk (0-10 for alcohol), moderate risk (11-26 for alcohol) or high risk (27 or higher for alcohol). The score range is 0-39. Higher score worse risk.
Time Frame: Baseline, 30 days, 60 days, 90 days, 180 days
Population: Restricted to participants who reported alcohol use at baseline. This outcome measures reduction in existing alcohol use among current users. Non-users were excluded as the intervention targets harm reduction rather than prevention of initiation.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | New Hope (NH) | Elders' Resiliency (ER) | Control Condition | New Hope (NH), Elders' Resiliency (ER), Case Management (CM)
Number analyzed (Participants) | 36 | 46 | 40 | 38
score on a scale
  Baseline | 19 [14.5 to 25.5] | 15 [8 to 23] | 18 [10 to 27] | 12 [2 to 18]
  30 Days: number analyzed (Participants) | 9 | 31 | 35 | 24
  30 Days | 5 [5 to 15] | 21 [10 to 26] | 21.5 [12 to 27] | 10 [5 to 22]
  60 Days: number analyzed (Participants) | 14 | 30 | 33 | 23
  60 Days | 9 [5 to 23] | 14 [8 to 28] | 15 [7 to 27] | 7.5 [3.5 to 11]
  90 Days: number analyzed (Participants) | 18 | 18 | 25 | 18
  90 Days | 6.5 [2 to 20] | 10.5 [5 to 17] | 20 [9 to 22] | 11 [3 to 21]
  180 Days: number analyzed (Participants) | 21 | 26 | 34 | 26
  180 Days | 20 [9 to 26] | 15 [5 to 23] | 11 [6 to 20] | 8 [5 to 13]

6. Primary Outcome: Suicide Ideation Questionnaire (SIQ)
Description: The SIQ for adults (ages >14; 27 items) and SIQ-Junior for youth (ages ≤14; 13 items). Both measure frequency of suicidal thoughts on a 7-point Likert scale (0=Never to 6=Almost Every Day). Raw scores range from 0-162 (SIQ) and 0-78 (SIQ-JR); higher raw scores indicate greater suicidal ideation. Raw scores of ≥30 on the SIQ and ≥23 on the SIQ-JR indicate clinically severe suicidal ideation.
  To create comparable scores across age groups, raw scores were converted to z-scores based on the study sample's baseline distribution, calculated separately for adults and youth using their respective scale versions. A constant of 10 was added to all z-scores to facilitate interpretation.
  Interpretation of Z-scores:
  * Each unit change represents one standard deviation from the sample
  * Z-scores >10 indicate above-average suicidal ideation (worse outcome)
  * Z-scores <10 indicate below-average suicidal ideation (better outcome) A Z-score of 0 represents the population mean
Time Frame: Baseline, 30 days, 60 days, 90 days, 180 days
Population: Participants with data collected
Measure: Median (Inter-Quartile Range); unit: Z-score
Arm/Group | New Hope (NH) | Elders' Resiliency (ER) | Control Condition | New Hope (NH), Elders' Resiliency (ER), Case Management (CM)
Number analyzed (Participants) | 71 | 68 | 80 | 65
Z-score
  Baseline | 10.2 [9.5 to 11.7] | 10 [9.3 to 10.7] | 10.1 [9.7 to 11.1] | 10.1 [9.4 to 11.4]
  30 Days: number analyzed (Participants) | 30 | 55 | 63 | 44
  30 Days | 9.9 [9.2 to 10.3] | 9.8 [9.2 to 10.2] | 9.9 [9.4 to 10.8] | 9.5 [9.2 to 10.1]
  60 Days: number analyzed (Participants) | 43 | 57 | 57 | 49
  60 Days | 9.6 [9.2 to 10.2] | 9.5 [9.2 to 10.1] | 9.7 [9.3 to 10.1] | 9.3 [9.2 to 10.1]
  90 Days: number analyzed (Participants) | 39 | 37 | 63 | 42
  90 Days | 9.5 [9.2 to 10.1] | 9.5 [9.2 to 9.7] | 9.8 [9.2 to 10.1] | 9.5 [9.2 to 10.0]
  180 Days: number analyzed (Participants) | 52 | 52 | 70 | 57
  180 Days | 9.4 [9.2 to 10.0] | 9.9 [9.3 to 10.3] | 9.3 [9.2 to 9.7] | 9.4 [9.2 to 10.1]

7. Primary Outcome: The Resiliency Scales
Description: Resilience Scales for Children and Adolescents (RSCA), adapted and validated with community input. The RSCA measures 3 domains of resilience using a 4-point Likert scale (0=Not at All, 1=A little bit, 2=A medium amount, 3=A lot):
  * Sense of Mastery: 20 items assessing self-efficacy and control (range: 0-60; higher better)
  * Sense of Relatedness: 18 items assessing trust and support from relationships (range: 0-54; higher better)
  * Emotional Reactivity: 24 items assessing vulnerability to stress and negative emotions (range: 0-72; lower better)
    1. Items are summed within each subscale
    2. Mastery and Relatedness subscales are summed to create a Resource Index (range: 0-114)
    3. The Total Resilience Score is calculated as: Resource Index minus Emotional Reactivity Total Resilience Score Range: -72 to 114
  Interpretation:
  * Higher scores indicate greater resilience (better outcome)
  * Better scores reflect more personal and relational resources combined with lower emotional vulnerab
Time Frame: Baseline, 30 days, 60 days, 90 days, 180 days
Population: Participants with data collected
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | New Hope (NH) | Elders' Resiliency (ER) | Control Condition | New Hope (NH), Elders' Resiliency (ER), Case Management (CM)
Number analyzed (Participants) | 71 | 68 | 80 | 65
Units on a scale
  Baseline | 31.7 (25.2) | 30.8 (21.5) | 33.3 (26.3) | 31.7 (22.7)
  30 Days: number analyzed (Participants) | 30 | 55 | 63 | 44
  30 Days | 43.9 (27.7) | 25.6 (26.9) | 33.8 (28) | 33.9 (28.6)
  60 Days: number analyzed (Participants) | 43 | 57 | 57 | 49
  60 Days | 46.2 (24.1) | 35.2 (25.1) | 39.4 (23.6) | 36.4 (30.8)
  90 Days: number analyzed (Participants) | 39 | 37 | 63 | 42
  90 Days | 40.9 (28.1) | 27.4 (19.7) | 39.8 (26) | 41.9 (29.8)
  180 Days: number analyzed (Participants) | 52 | 52 | 70 | 57
  180 Days | 50.5 (24.2) | 30.5 (26.7) | 43.4 (27.7) | 42.3 (29.9)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, 6 months
Description: AEs could be reported to study staff during study visits with participants, in alerts from the ER or hospital, or alerts from participant or family members outside of study visits. AEs were then recorded by the study team and reported to IRB and sponsor as required.
Arm/Group | New Hope (NH) | Elders' Resiliency (ER) | New Hope (NH), Elders' Resiliency (ER), Case Management (CM) | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/68 | 0/65 | 0/80
Serious Adverse Events (participants affected / at risk) | 15/71 | 10/68 | 10/65 | 15/80
Other Adverse Events (participants affected / at risk) | 5/71 | 1/68 | 0/65 | 4/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Hope (NH) (N=71) | Elders' Resiliency (ER) (N=68) | New Hope (NH), Elders' Resiliency (ER), Case Management (CM) (N=65) | Control Condition (N=80)
ER Treatment for Suicide Ideation (Psychiatric disorders) | 7 | 6 | 5 | 7 — Participant seen in ER for SI, discharged home
In-patient treatment for SI (Psychiatric disorders) | 8 | 4 | 5 | 8 — Participant sent to in-patient treatment for SI
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Hope (NH) (N=71) | Elders' Resiliency (ER) (N=68) | New Hope (NH), Elders' Resiliency (ER), Case Management (CM) (N=65) | Control Condition (N=80)
Incarceration (General disorders) | 3 | 0 | 0 | 3 — Participant incarcerated
Other hospitalization (General disorders) | 0 | 1 | 0 | 1 — not-mental health related visit to ER or hospital
Expelled from school (General disorders) | 1 | 0 | 0 | 0
Sexual abuse (General disorders) | 1 | 0 | 0 | 0 — abuse/assault of participant, reported to study team and reported to BIA

LIMITATIONS AND CAVEATS:
Study limitations include constraints on generalizability, as our sample was predominantly female (73%) and conducted within a single Tribal Nation, limiting the generalizability of our findings. The study design did not permit isolation of the specific effects of case management alone; this was intentional and ethically necessary. The pandemic fundamentally compromised ERC implementation, and the intervention's full potential should be evaluated in a future study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT03543865/Prot_SAP_000.pdf
  • Informed Consent Form: Adult Informed Consent (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT03543865/ICF_001.pdf
  • Informed Consent Form: Parent Informed Consent (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT03543865/ICF_002.pdf
  • Informed Consent Form: Youth Informed Assent (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT03543865/ICF_003.pdf